CLINICAL TRIAL: NCT07061600
Title: Mental Health Literacy in the Digital Age: Assessing the Efficacy and Acceptance of a Social Media Intervention for Adolescent Depression With a Randomized Controlled Trial
Brief Title: Enhancing Depression Literacy and Reducing Stigma in Adolescents Through Social Media
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Prof. Otto Beisheim Foundation (Other)
Responsible Party: Principal Investigator, Ellen Greimel, Working group leader, LMU Klinikum
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 25-0085
Record Dates: First submitted 2025-06-26; First posted 2025-07-11 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Depressive Disorder; Depression - Major Depressive Disorder; Depression in Adolescence
Keywords: depression; social media; adolescents; depression literacy; stigma; help-seeking; psychoeducation; ecological momentary assessment
MeSH Terms: conditions — Depressive Disorder; Depression; Social Stigma

STUDY DESIGN:
Intervention Model Description: After the recruitment phase, the participants are randomly assigned to either the experimental group (EG), which receives "ich bin alles" Instagram content, or the control group (CG) before the start of the study. The control group receives content from an Instagram profile in the field of education that is not related to mental health issues (https://www.instagram.com/terrax/?hl=de). Randomisation is carried out using 1:1 randomisation, stratified by age (< 16 years vs. ≥ 16 years) and gender. With the exception of one team member, who will be responsible for the administration and randomisation of participants and will not be involved in the statistical analyses, participants and staff will be blind to allocation.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: With the exception of one team member, who will be responsible for the administration and randomisation of participants and will not be involved in the statistical analyses, participants and staff will be blind to allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "ich bin alles" (Instagram profile) (Experimental): The experimental group is encouraged to follow the "ich bin alles" Instagram account closely and to view the posted information material regularly over the period of 4 weeks.
  Interventions: Behavioral: "ich bin alles"
- Control Group (Active Comparator): The active control group is asked to follow an Instagram profile that provides educational content produced by a public broadcaster. The educational content is not related to mental health issues (https://www.instagram.com/terrax/?hl=de).
  Interventions: Behavioral: Instagram profile that provides educational content

INTERVENTIONS:
Behavioral: "ich bin alles" — The web-based information platform "ich bin alles" (www-ich-bin-alles.de) on depression and mental health in youth as well as its Social Media channels were developed by the Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy of the LMU Munich Hospital together with the Prof. Otto Beisheim Foundation. It is aimed at youth with depression, healthy youth, and their parents. The project focuses on education, prevention, low-threshold support, and destigmatisation through the transfer of evidence-based knowledge and hands-on supportive materials. Information material on Instagram is posted four times a week in the form of a post, a longer explanatory video and two reels (i.e. short videos with overlays of text and music). All content is evidence-based information created by the research team and is primarily based on the "ich bin alles" page.
  Arms: "ich bin alles" (Instagram profile)
Behavioral: Instagram profile that provides educational content — The participants of the control group asked to follow an Instagram profile that provides educational content produced by a public broadcaster (https://www.instagram.com/terrax/) and is not dedicated to the topic of mental health. This channel also posts several times a week and provides educational or informational content.
  Other Names: terrax
  Arms: Control Group

SUMMARY:
Depression is a highly common mental disorder that often begins in adolescence. Despite its high burden and negative consequences, few young people seek professional help due to, e.g., low mental health literacy and fear of stigma. Since adolescents frequently seek health information online and use social media daily, the project "ich bin alles" (English: "I am everything"; www.ich-bin-alles.de) was launched to provide easily accessible, age-appropriate, and evidence-based information about depression and mental health via digital platforms including a website and social media channels (e.g., Instagram). This study aims to evaluate the effectiveness of the "ich bin alles"- Instagram channel in improving depression literacy, reducing stigma, and encouraging help-seeking behavior, as well as assessing user acceptance and content reception.

DETAILED DESCRIPTION:
Depression is one of the most common mental disorders worldwide, with a prevalence of up to 7.5% in children and adolescents. In connection with the COVID-19 pandemic, a meta-analysis found an increase in clinically relevant depressive symptoms to 25.2% in children and adolescents. At the same time, adolescents who experience mental health crises are reluctant to seek help and only 12% of adolescents with clinically relevant depressive symptoms seek professional treatment. The main barriers for young people to seek professional help include low knowledge of mental disorders/low mental health literacy and social factors such as the fear of stigmatization. Mental health literacy (MHL) is defined as "how to prevent mental disorders, recognition of when a disorder is developing, knowledge of help-seeking options and treatment available, knowledge of effective self-help strategies for milder problems, and first aid skills to support others who are affected by mental health problems". It has been found that increased depression literacy can reduce depressive symptoms in adults and improve help-seeking for depression.

Stigma in the context of mental health is a multidimensional concept that encompasses several domains. For many people living with mental illness, stigma is a significant contributor to a wide range of negative outcomes, including delayed help-seeking, hopelessness, diminished self-esteem, reduced quality of life and poorer clinical outcomes. Many of these negative effects have also been found in young people with mental health problems. Therefore, improving MHL and reducing the stigmatization of mental illness are two important starting points that can serve as targets for interventions. Improved MHL goes hand in hand with better knowledge about seeking help and less stigmatization of mental illness.

The vast majority of adolescents in western countries, such as the US and Germany, have access to digital devices, such as smartphones, 97% of young people in the U.S. (13-17 years) state that they use social media and 45% say that they are online almost all the time. Along with this, young people are more likely to ask health questions, including mental health questions, online than through other channels. However, to date, few digital psychoeducational interventions for depression in adolescents have been developed and evaluated. In order to meet this need for action in a contemporary manner that attracts youth, the web-based project "ich bin alles" (English: "I am everything"; www.ich-bin-alles.de) was launched in September 2021 with an associated social media presence. The "ich bin alles" project provides comprehensive evidence-based and age-appropriate information on depression and mental health in youth via social media (such as Instagram).

The aim of this study is to investigate in a randomized controlled trial whether educating adolescents via Instagram is an effective and accepted method to inform about depression and mental health. In more detail, the effects of targeted communication of content via Instagram on (1) information regarding the appearance, causes, and development of depression, (2) stigma towards depression, and (3) help-seeking behaviour are investigated. It is examined whether this communication of information leads to an increase in depression literacy, a reduction in stigma, and an increase in the intention to seek help and whether these changes are maintained over three months. Furthermore, the acceptance of the content will be investigated.

In this study, participants will be randomly assigned to either an experimental group (EG) or an active control group (CG). Participants assigned to the EG will be asked to regularly consume "ich bin alles" Instagram content over the period of four weeks. The CG will be asked to regularly view content from an Instagram channel from the field of education created by a public broadcaster (https://www.instagram.com/terrax/) over the same time period. Before the reception of the content (pre), after four weeks (post), and at a three months follow-up, participants will fill out questionnaires via an app ("m-Path"), with each assessment lasting approx. 30 minutes. At each assessment point, participants simultaneously receive a push notification via the app to complete the questionnaire. The pre-assessment is intended to check the eligibility criteria and record demographic data such as gender, highest educational qualification, and current employment/education status. The primary outcome measures (depression literacy, intention to seek help, stigma) are assessed at pre, post, and follow-up. After 4 weeks, the post assessment will take place, during which acceptance is also tested in addition to the primary outcome measures. After another 3 months, the follow-up assessment is scheduled. During the four-week intervention period, Ecological Momentary Assessment will be used to ask adolescents a few short questions every day about their mood and their use of the Instagram channel via the m-Path app.

ELIGIBILITY:
Inclusion Criteria:

* Ownership of an Instagram account
* Regular use of Instagram

Exclusion Criteria:

* No exclusion citeria

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 170 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
Depression Literacy | Pre-test (week 0), post-test (week 4), follow-up (week 16)
  Assessed with an adapted version of the German version of the Adolescent Depression Knowledge Questionnaire and the Depression Literacy Scale German
Stigma | Pre-test (week 0), post-test (week 4), follow-up (week 16)
  Stigma - Assessed with the German version of the Self Stigma of Depression Scale and adapted Version of the Peer mental health stigmatization scale
Intention to seek help | Pre-test (week 0), post-test (week 4), follow-up (week 16)
  Assessed using the German version of the Attitudes Toward Seeking Professional Psychological Help Scale - Short Form
Mental Health | Pre-test (week 0), post-test (week 4), follow-up (week 16)
  Assessed with the Depression Screener for Teenagers and the Perceived Stress Scale
Visual Aesthetics | post-test (week 4)
  Assessed via an adapted version of the Visual Aesthetics of Website Inventory - Short
Intentions to act | post-test (week 4)
  Assessed via an adapted version of the Scale assessing the intention to revisit the website
Overall impression | post-test (week 4)
  assessed via a single item based on Thielsch

SECONDARY OUTCOMES:
Ecological Momentary Assessment (Control function and mood changes) | every day between Pre-test (week 0) and post-test (week 4)
  Changes in mood and consumption of Instagram profiles over the period of the intervention through daily surveys using specially created items

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Schulte-Körne, Prof. Dr., Principal Investigator — Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy, Hospital of the Ludwig-Maximilians-University (LMU) Munich
Locations (1):
- Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy, Hospital of the Ludwig-Maximilians-University (LMU) Munich, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No
The data collected in this study include sensitive details about participants, such as various sociodemographic characteristics. Publicly sharing the raw dataset could risk revealing individual identities, thereby violating ethical standards related to participant confidentiality. As a result, the raw data will not be publicly released. However, detailed descriptions of the methodology, materials used, and sample characteristics will be provided within the article and supplementary materials. The intervention is also publicly accessible in German on the "ich bin alles" - Instagram channel. Aggregated data and additional supporting materials may be shared upon request (contact: sara.kaubisch@med.uni-muenchen.de).

REFERENCES:
- See also: Related Info — https://www.instagram.com/ich.bin.alles/